CLINICAL TRIAL: NCT05138510
Title: Sexuality and Breast Cancer: Developing Appropriate Education for Women Going Through Treatment
Brief Title: Sexual Health in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1789.cc; NCI-2021-10894 (Other: CTRP)
Record Dates: First submitted 2021-10-26; First posted 2021-12-01 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Stage 0: Ductal carcinoma in situ. Timing: start of endocrine therapy
  Interventions: Behavioral: Focus Group
- Stages I-III Surgery first: Invasive cancer. Surgery first Timing: start of endocrine therapy
  Interventions: Behavioral: Focus Group
- Stages I-III, neoadjuvant chemotherapy first: Invasive cancer. Neoadjuvant chemotherapy first Timing: during neoadjuvant chemotherapy
  Interventions: Behavioral: Focus Group
- Stage IV: Metastatic cancer, chemotherapy only, no invasive surgery Timing: 2 months into treatment
  Interventions: Behavioral: Focus Group
- Survivors: Timing: any time
  Interventions: Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Focus Group — Providers with extensive training and expertise in the subject will lead the virtual focus groups over Zoom using a semi-structured guide. Topics will focus on education received from the health care team, information received from outside sources, and patient recommendations on the type and timing of information preferred.
  We will create an analytic report based on the focus group findings, which will be used to inform the development of educational material.
  Sexual well-being is currently measured longitudinally on a 0-100 point scale as a component of a validated patient-reported outcome measures (PROM) survey (BREAST-Q) distributed to all breast cancer patients. These scores will be analyzed in patients with and without educational interventions for comparison.

SUMMARY:
In the present study, we propose a mixed methods approach to characterize and address the sexual health needs among women with breast cancer at the time of diagnosis and throughout treatment.

DETAILED DESCRIPTION:
In the present study, we propose a mixed methods approach to characterize and address the sexual health needs among women with breast cancer at the time of diagnosis and throughout treatment. The objectives are as follows:

1. To characterize the sexual well-being of women longitudinally throughout the continuum of care, from initial diagnosis into survivorship.

   We predict that treatment will adversely affect sexual well-being, and that patient factors, clinical factors, and treatment choices will influence changes in sexual well-being.
2. To identify gaps is sexual health education provided at the time of diagnosis or during treatment and to determine the appropriate timing of sexual health education delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ductal carcinoma in situ or invasive breast cancer, seen in the breast center between 09/01/2019 to present, will potentially be recruited to participate.

Exclusion Criteria:

* Patients less than 18 years of age and those with non-cancer diagnoses or prior history of breast cancer will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All patients diagnosed with ductal carcinoma in situ or invasive breast cancer, seen in the breast center between 9/1/2019 to present, will potentially be recruited to participate. Patients less than 18 years of age and those with non-cancer diagnoses or prior history of breast cancer will be excluded.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Determine changes in sexual well-being for women with breast cancer | 1 year
  Determine changes in sexual well-being throughout the course of breast cancer treatment, pre- and post-implementation of developed educational materials using the Sexual Health Among Women Receiving Breast Cancer Treatment Survey
Determine educational resources currently used for sexual health information | 1 year
  Determine patients' self reported list of educational media received regarding sexual health during breast cancer treatment using the PROM survey (BREAST-Q)
Determine educational resources currently used for sexual health information | 1 year
  Determine patients' self reported list of educational media received regarding sexual health during breast cancer treatment using the Sexual Health Among Women Receiving Breast Cancer Treatment Survey
Determine patients preferred type of education for sexual health | 1 year
  Determine the patients preferred type and timing of educational interventions for sexual health using the Sexual Health Among Women Receiving Breast Cancer Treatment Survey

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tevis, Principal Investigator — Colorado Research Center
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers. Individual Participant Data will be housed in a deidentified format in the secure, encrypted REDCap database of the University of Colorado School od Medicine.